CLINICAL TRIAL: NCT06846320
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Fixed-Dose Study to Evaluate the Efficacy, Safety, and Tolerability of ABBV-932 as an Adjunct to Antidepressant Therapies in the Treatment of Subjects With Generalized Anxiety Disorder Who Have Had an Inadequate Response to Antidepressant Therapies
Brief Title: Study to Assess Adverse Events and Change in Disease Activity When Oral ABBV-932 is Added to Antidepressant Therapies in Adult Participants With Generalized Anxiety Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M25-099
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Generalized Anxiety Disorder (GAD)
Keywords: LEGATO - (GAD); Generalized Anxiety Disorder (GAD); ABBV-932
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- ABBV-932 Dose A (Experimental): Participants will receive ABBV-932 dose A in addition to prescribed antidepressant therapies (ADTs).
  Interventions: Drug: ABBV-932; Drug: Antidepressant Therapy (ADT)
- ABBV-932 Dose B (Experimental): Participants will receive ABBV-932 dose B in addition to prescribed antidepressant therapies (ADTs).
  Interventions: Drug: ABBV-932; Drug: Antidepressant Therapy (ADT)
- Placebo for ABBV-932 (Placebo Comparator): Participants will receive placebo for ABBV-932 in addition to prescribed antidepressant therapies (ADTs).
  Interventions: Drug: Placebo for ABBV-932; Drug: Antidepressant Therapy (ADT)

INTERVENTIONS:
Drug: ABBV-932 — Oral Capsule
  Arms: ABBV-932 Dose A; ABBV-932 Dose B
Drug: Placebo for ABBV-932 — Oral Capsule
  Arms: Placebo for ABBV-932
Drug: Antidepressant Therapy (ADT) — Standard of care

SUMMARY:
Generalized anxiety disorder (GAD) is usually treated with antidepressant therapy (ADT); however, sometimes ADTs alone are not enough to adequately treat GAD. The purpose of this study is to assess how safe and effective ABBV-932 is when added to the antidepressant therapies in adult participants with GAD who have had an inadequate response ADTs.

ABBV-932 is an investigational drug being developed for the adjunctive treatment of GAD. Participants will be randomly assigned to receive ABBV-932 or Placebo in addition to their currently prescribed ADTs. There is 1 in 3 chance of participants assigned to Placebo. Approximately 315 adult participants with GAD and inadequate response to ADTs will be enrolled in approximately 50 sites in the United States and Puerto Rico.

Participants will receive oral capsules of ABBV-932 or matching placebo in addition to their prescribed ADT for 6 weeks and then will be followed for an additional 4 week follow-up period.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Meet Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision (DSM-5-TR) criteria for generalized anxiety disorder (GAD) confirmed by the Mini International Neuropsychiatric Interview (MINI).
* Currently taking one of the Food and Drug Administration (FDA) approved antidepressant therapies (ADT) for GAD (i.e., escitalopram, paroxetine, duloxetine, or venlafaxine ER) with an inadequate response to an adequate dose (per label) and duration (>= 8 weeks) as verified by a baseline Hamilton Anxiety Rating Scale (HAM-A) total score >= 20 and Clinical Global Impression of Severity Scale (CGI-S GAD) >= 4.

Exclusion Criteria:

* Have a Montgomery-Åsberg Depression Rating Scale (MADRS) score >= 20.
* New diagnosis or exacerbation of major depression in the last 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to approximately 10 weeks
  An AE is defined as any untoward medical occurrence in which a participant is administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.
Change from Baseline in the Hamilton Anxiety Scale (HAM-A) Total Score | Up to approximately 6 weeks
  The HAM-A is a 14-item, clinician-reported measure used to quantify and categorize the participant's anxiety over the past week. Items are rated on a 5-point Likert rating scale. The HAM-A total score ranges from 0 to 56, with higher scores indicating greater anxiety severity.

SECONDARY OUTCOMES:
Change from Baseline in Penn State Worry Questionnaire-10 (PSWQ-10) Total Score | Up to approximately 6 weeks
  The PSWQ-10 is a 10-item, participant-reported measure of the tendency of an individual to worry, the excessiveness or intensity of worry, and the tendency for the worry to be generalized and not restricted to a small number of situations. Items are rated from 0 to 6 (0, never; 6, almost always). Total scores range from 0 to 60, with higher scores indicating greater worry.
Change from Baseline in Clinical Global Impression of Severity Scale (CGI-S) Generalized Anxiety Disorder (GAD) | Up to approximately 6 weeks
  The CGI-S GAD is a single, clinician-reported item that measures the clinician's impression of a participant's current anxiety severity considering their total clinical experience with the participant population. The measure uses a 5-point Likert rating scale, with higher scores indicating greater anxiety severity.
Change from Baseline in the Hamilton Anxiety Scale (HAM-A) Total Score | Up to approximately 4 weeks
  The HAM-A is a 14-item, clinician-reported measure used to quantify and categorize the participant's anxiety over the past week. Items are rated on a 5-point Likert rating scale. The HAM-A total score ranges from 0 to 56, with higher scores indicating greater anxiety severity.
Change From Baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score | Up to approximately 6 weeks
  The MADRS is a 10-item, clinician-rated scale that evaluates the participant's depressive symptomatology during the past week. Participants are rated on items assessing feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty in concentration, and lack of interest. Each item is scored on a 7-point scale with a score of 0 reflecting no symptoms and a score of 6 reflecting symptoms of maximum severity.
Percentage of Participants in Remission | Up to approximately 6 weeks
  Remission is defined as HAM-A total score <=7.
Percentage of Participants with HAM-A Response | Up to approximately 6 weeks
  HAM-A response is defined as >= 50% reduction from baseline in HAM-A total score
Percentage of Participants with Clinical Global Impression of Change (CGI-C) GAD Responder Status of "Much Better" or "Moderately Better" | Up to approximately 6 weeks
  The CGI-C GAD is a clinician-rated scale that measures the overall change in a participant's GAD symptoms since initial receipt of the study medication. The participant is rated on a 7-point Likert scale ranging from "Much better" (1) to "Much worse" (7).
Change from Baseline in Patient Global Impression of Severity Scale (PGI-S) Generalized Anxiety Disorder (GAD) | Up to approximately 6 weeks
  The PGI-S GAD is a single, patient-reported item that assesses the subject's perceived level of GAD symptoms over the past 7 days. The measure uses a 5-point Likert rating scale with responses ranging from "no symptoms" (1) to "very severe" (5), with higher scores indicating greater severity of GAD symptoms.
Percentage of Participants with Patient Global Impression of Change Scale (PGI-C) Generalized Anxiety Disorder (GAD) Responder Status of "Much Better" or "Moderately Better" | Up to approximately 6 weeks
  The PGI-C GAD is a single, patient-reported item that assesses the subject's perceived overall change in their GAD symptoms since they started taking the study medication. The measure uses a 7-point Likert rating scale with responses ranging from "much better" (1) to "much worse" (7). Higher scores indicate worse GAD symptoms
Change from Baseline in Patient Global Impression of Severity Scale (PGI-S) Worry | Up to approximately 6 weeks
  The PGI-C Worry is a single, patient-reported item that assesses the subject's perceived overall change in their worry since they started taking the study medication. The measure uses a 7-point Likert rating scale with responses ranging from "much less worried" (1) to "much more worried" (7). Higher scores indicate more worry.
Percentage of Participants with Patient Global Impression of Change Scale (PGI-C) Worry Responder Status of "Much Better" or "Moderately Better" | Up to approximately 6 weeks
  The PGI-C Worry is a single, patient-reported item that assesses the subject's perceived overall change in their worry since they started taking the study medication. The measure uses a 7-point Likert rating scale with responses ranging from "much less worried" (1) to "much more worried" (7). Higher scores indicate more worry.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (52):
- United States (49):
  - University of Alabama - Huntsville Regional Medical Campus /ID# 267818, Huntsville, Alabama
  - Ima Clinical Research Phoenix (Alea) /ID# 275737, Phoenix, Arizona
  - Noble Clinical Research /ID# 267952, Tucson, Arizona
  - Advanced Research Center /ID# 267874, Anaheim, California
  - Axiom Research /ID# 267814, Colton, California
  - Sun Valley Research Center /ID# 267864, Imperial, California
  - Synergy San Diego /ID# 267879, Lemon Grove, California
  - Alliance for Research Alliance for Wellness /ID# 267911, Long Beach, California
  - NRC Research Institute DTLA /ID# 267832, Los Angeles, California
  - Excell Research /ID# 267918, Oceanside, California
  - Viking Clinical Research Center - Temecula /ID# 268598, Temecula, California
  - Sunwise Clinical Research /ID# 267863, Walnut Creek, California
  - Connecticut Clinical Research - Cromwell /ID# 271241, Cromwell, Connecticut
  - Cns Healthcare - Jacksonville /ID# 268588, Jacksonville, Florida
  - Accel Research Sites Network - St. Pete /ID# 267821, Largo, Florida
  - K2 Medical Research, LLC /ID# 267841, Maitland, Florida
  - GMI Florida - Central Miami Medical Institute /ID# 267839, Miami, Florida
  - Allied Biomedical Res Inst Inc /ID# 267813, Miami, Florida
  - Apg Research /ID# 271707, Orlando, Florida
  - Psych Atlanta /ID# 267878, Marietta, Georgia
  - iResearch Savannah /ID# 267865, Savannah, Georgia
  - University of Chicago Medical Center /ID# 275131, Chicago, Illinois
  - Collective Medical Research /ID# 272015, Overland Park, Kansas
  - CenExel /ID# 267853, Gaithersburg, Maryland
  - Elixia, LLC /ID# 267815, Springfield, Massachusetts
  - Psychiatric Care And Research Center /ID# 271701, O'Fallon, Missouri
  - St. Charles Psychiatric Associates /ID# 271202, Saint Charles, Missouri
  - Arch Clinical Trials /ID# 267851, St Louis, Missouri
  - Ima Clinical Research Las Vegas (Altea) /ID# 275731, Las Vegas, Nevada
  - Duplicate_Oasis Clinical Research, LLC /ID# 267953, Las Vegas, Nevada
  - Princeton Medical Institute /ID# 267877, Princeton, New Jersey
  - Bio Behavioral Health /ID# 267919, Toms River, New Jersey
  - Integrative Clinical Trials /ID# 279519, Brooklyn, New York
  - New Hope Clinical Research - Inpatient unit /ID# 267810, Charlotte, North Carolina
  - Quest Therapeutics of Avon /ID# 267829, Avon Lake, Ohio
  - University Of Cincinnati Medical Center /ID# 271704, Cincinnati, Ohio
  - The Ohio State University /ID# 267924, Columbus, Ohio
  - Sooner Clinical Research /ID# 267881, Oklahoma City, Oklahoma
  - Lehigh Center for Clinical Research /ID# 267908, Allentown, Pennsylvania
  - Suburban Research Associates /ID# 267868, West Chester, Pennsylvania
  - Coastal Carolina Research Center, LLC /ID# 267826, Charleston, South Carolina
  - Psychiatric Consultants - Franklin /ID# 275133, Franklin, Tennessee
  - FutureSearch Trials of Dallas /ID# 267870, Dallas, Texas
  - Relaro Medical Trials /ID# 270241, Dallas, Texas
  - Perceptive Pharma Research /ID# 267836, Richmond, Texas
  - Family Psychiatry Of The Woodlands /ID# 275173, The Woodlands, Texas
  - Grayline Research Center /ID# 267811, Wichita Falls, Texas
  - Northwest Clinical Research Center /ID# 267916, Bellevue, Washington
  - Core Clinical Research /ID# 270058, Everett, Washington
- Puerto Rico (3):
  - INSPIRA Clinical Research /ID# 267822, San Juan
  - Instituto De Neurologia Dra. Ivonne Fraga, Psc /ID# 267793, San Juan
  - BDH Research /ID# 267787, San Juan

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-099